CLINICAL TRIAL: NCT00219297
Title: An Open-label, Multi-center, Phase II Study to Evaluate the Activity of Patupilone (EPO906), in the Treatment of Recurrent or Progressive Brain Metastases in Patients With Non-small Cell Lung Cancer.
Brief Title: Study of Patupilone in Patients With Brain Metastasis From Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2227
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Brain Metastasis; Non-small Cell Lung Cancer
Keywords: EPO; EPO906; Brain cancer; Brain metastasis; Lung cancer; Lung metastasis; Brain metastasis from non-small cell lung cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — epothilone B

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Patupilone

INTERVENTIONS:
Drug: Patupilone

SUMMARY:
The study objective is to evaluate the safety and efficacy of patupilone with respect to early progression and response of patients with non-small cell lung cancer (NSCLC) metastatic to the brain, who have progressed after chemotherapy, surgery and/or radiation.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) performance status of 0, 1 or 2 (corresponding to Karnofsky performance status of 50 or better)
* Patients with radiologically proven (by gadolinium-enhanced [Gd-] magnetic resonance imaging [MRI]) parenchymal brain metastases from histologically confirmed non-small cell lung cancer (the primary disease may be quiescent). Gd-MRI must be performed within 2 weeks of study entry.
* Patients should have at least one bidimensionally measurable intracranial lesion of a minimum of 2 cm as defined by Gd-MRI. If the patient has had previous radiation to the marker lesion(s), there must be evidence of residual disease > 2 cm or the lesion must have demonstrated progression since the radiation.
* Those patients progressing on radiotherapy must have a 25% increase in the size of the previously radiated intracranial lesion based on the Neuro-Oncology Criteria of Tumor Response for Central Nervous System (CNS) Tumors or appearance of new lesions.
* Patients must be controlled on medication and neurologically stable: stable on steroids and anticonvulsants for at least 2 weeks prior to obtaining the baseline Gd-MRI of the brain, and/or at least 2 weeks prior to beginning study treatment.
* Female patients must have a negative serum pregnancy test at screening. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal.)
* All patients of reproductive potential must agree to use an effective method of contraception during the study and for three months following termination of treatment.
* Written informed consent must be obtained.

Exclusion Criteria:

* Clinical evidence of leptomeningeal disease
* Patients with extracranial disease in more than 3 organ sites including the primary tumor.
* Patients who have received any investigational compound within the past 28 days or who are planning to receive other investigational drugs while participating in the study
* Prior administration of epothilone(s)
* Patients with peripheral neuropathy > grade 1
* Patients with unresolved diarrhea within the last 7 days before treatment.
* Patients receiving known diarrheogenic agents must stop treatment with these agents prior to enrollment in the study.
* Radiotherapy < 3 weeks prior to study entry
* Prior intracranial surgery < 3 weeks prior to study entry; patient must have recovered from surgery prior to study entry.
* Chemotherapy < 3 weeks prior to study entry; < 6 weeks from prior nitrosoureas.
* Severe cardiac insufficiency (New York Heart Association [NYHA] III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease
* Radiotherapy not permitted while on study. Exception: palliative radiotherapy of metastasis in extremities is allowed, but such lesions cannot be used as target or non-target lesions.
* Patients receiving hematopoietic growth factors except for erythropoietin
* Patients taking Coumadin® or other agents containing warfarin, with the exception of low dose Coumadin® (1 mg or less daily) administered prophylactically for maintenance of in-dwelling lines or ports

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-11-16 (Actual); Primary Completion 2010-06-24 (Actual); Study Completion 2010-06-24 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST) | throughout the study

SECONDARY OUTCOMES:
Time to progression of the brain metastases | throughout the study
Pharmacokinetics (PK) of patupilone in blood | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - University of California Davis Cancer Center UC Davis Cancer (3), Sacramento, California
  - Dana Farber Cancer Institute SC, Boston, Massachusetts
  - Wayne State University/Wertz Clinical Cancer Center Div. of Hematology/Oncology, Detroit, Michigan
  - St Louis University Cancer Center, St Louis, Missouri
  - Washington University School of Medicine-Siteman Cancer Ctr, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center Oncology, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center New York Presbyterian, New York, New York
  - Duke University Medical Center Dept. of DUMC (3), Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5726